CLINICAL TRIAL: NCT02252549
Title: The SPIES Non-Muscle-Invasive Bladder Cancer Study - A Multicenter Randomized Controlled Study; A Multicenter International Randomized Controlled Study to Compare the Outcome Using the Storz Professional Image Enhancement System (SPIES) Versus White Light Imaging (WLI) During TURB of Non-Muscle-Invasive Bladder Cancer (NMIBC).
Brief Title: An International Randomized Study to Compare SPIES Versus WLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL50451.018.14
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): SPIES+WLI assisted TURB
  Interventions: Device: SPIES+WLI assisted TURB
- B (Active Comparator): WLI assisted TURB
  Interventions: Device: WLI assisted TURB

INTERVENTIONS:
Device: SPIES+WLI assisted TURB
  Arms: A
Device: WLI assisted TURB
  Arms: B

SUMMARY:
This study is a multicenter randomized controlled trial in which the efficacy between SPIES assisted and WLI assisted TURB are compared. Subjects in the experimental arm (Arm A) will undergo SPIES assisted TURB, whereas subjects in the control arm (Arm B) will receive treatment with WLI assisted TURB only. Baseline characteristics will be recorded, as well as short and long-term follow up.

DETAILED DESCRIPTION:
This study is a multicenter randomized controlled trial in which the recurrence rates of cancer between SPIES assisted and WLI assisted TURB are compared. Randomization is stratified by tumor multiplicity (single or multiple), tumor status (primary or recurrent) and macroscopic findings (papillary or flat, where CIS is scored as flat lesion). Patients randomized into the experimental arm (Arm A) will undergo SPIES and WLI assisted TURB, whereas the patients in the control arm (Arm B) will undergo WLI only assisted TURB. WLI is chosen as control, since it is considered the gold standard for detecting bladder tumors. Short and long term follow up will be recorded in order to evaluate the health gains for patients over a longer period. Perioperative (30 days) complications will be compared between the two treatment arms to evaluate the safety of SPIES.

ELIGIBILITY:
Inclusion Criteria:

* Has signed informed consent
* Is scheduled for treatment of a primary or recurrent NMIBC
* Is aged 18 years or older
* Has or has had no tumors in the upper urinary tract
* Has had no previous irradiation of the pelvis

Exclusion Criteria:

* Gross haematuria at the time of TURB (i.e. heavy bladder bleeding resulting in marked amounts of blood in the urine which may interfere with cystoscopy)
* Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days
* Pregnancy or breast-feeding (all women of child-bearing potential must document a negative serum or urine pregnancy test at screening and are suggested to use the contraceptive pill or an intrauterine device (IUD) during the treatments and for at least one months thereafter)
* Conditions associated with a risk of poor protocol compliance
* Has had instillation therapy in the six months prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2015-04; Primary Completion 2020-04 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
To compare the recurrence rate of tumor at 12 months following SPIES assisted TURB (Arm A) with White Light Imaging only assisted TURB (Arm B) | 1 year

SECONDARY OUTCOMES:
1. To assess the recurrence rate of tumor at short and long term follow up (3 months and 3 years) after SPIES or WLI assisted TURB in patients with NMIBC. | 3 years
2. To assess the peri-operative morbidity (30 days) between SPIES and WLI assisted TURB by comparing the proportion of adverse events and using the Clavien-Dindo score. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean de la Rosette, Study Chair — Clinical Research Office of the Endourological Society

REFERENCES:
- [Derived] de la Rosette J, Martov A, Hurle R, Favre G, Mamoulakis C, Castanheira de Oliveira M, Stenzl A, Linares-Espinos E, Trelles Guzman CR, Gravas S, Knoll T, Boz MY, Herrmann T, Laguna P. Conventional white light imaging-assisted transurethral resection of bladder tumour (TURBT) versus IMAGE1S-assisted TURBT in non-muscle-invasive bladder cancer patients: trial protocol and 18 months results. World J Urol. 2022 Mar;40(3):727-738. doi: 10.1007/s00345-021-03866-4. Epub 2021 Nov 6. PMID 34741631